CLINICAL TRIAL: NCT06891937
Title: A Self-directed Positive Psychology Intervention for Individuals With Newly Diagnosed Multiple Sclerosis
Brief Title: Self-Directed Positive Psychology Intervention for Newly Diagnosed Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bonnie Ilene Glanz, Research Associate, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003100
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Positive psychology; Positive affect
MeSH Terms: conditions — Multiple Sclerosis | interventions — Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Subjects randomized to the intervention group will complete questionnaires at enrollment, Week 5 and Week 10. They will also complete 5 weeks of PP exercises, one exercise per week, during the intervention phase (weeks 1-5) of the study.
  Interventions: Behavioral: Positive psychology
- Waitlist Control (Placebo Comparator): Subjects randomized to the waitlist control group will complete study questionnaires at enrollment, Week 5 and Week 10. They will also complete 5 weeks of PP exercises, one exercise per week, during the extension phase (weeks 6-10) of the study.
  Interventions: Behavioral: Positive psychology

INTERVENTIONS:
Behavioral: Positive psychology — 5-week positive psychology intervention

SUMMARY:
The goal of this clinical trial is to learn whether positive psychology (PP) exercises such as writing a letter of gratitude or remembering a past success can help individuals with newly diagnosed multiple sclerosis (MS) to feel more hopeful, happy, and healthy. The main questions it aims to answer are:

* Is a five-week self-directed PP training intervention feasible and acceptable to individuals with newly diagnosed MS?
* Does the completion of a five-week self-directed PP training intervention improve positive affect, emotional function and health-related quality of life (HRQOL) in individuals with newly diagnosed MS?
* Are improvements in positive affect, emotional function and HRQOL maintained after the completion of the intervention?

Participants will be randomized to the intervention or waitlist control group. There will be an intervention phase (weeks 1-5) and an extension phase (weeks 6-10). All participants will complete questionnaires at enrollment, 5 weeks and 10 weeks. They will complete 5 weeks of self-directed PP training exercises, either during the intervention phase (intervention group) or extension phase (waitlist control group) of the study.

Researchers will compare participants in the intervention and waitlist control groups at the end of the intervention phase to see if there are improvements in positive affect, emotional function and HRQOL. For subjects in the intervention group who demonstrate improvement, researchers will determine if the benefit is maintained by comparing positive affect, emotional function and HRQOL at the completion of the intervention and extension phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS according to the McDonald 2017 diagnostic criteria
* Onset of disease within the last 2 years
* Ability to speak, read and write in English

Exclusion Criteria:

• Moderate or marked cognitive abnormalities identified by the treating neurologist during routine clinical visits that would preclude meaningful participation in the PP exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham MS Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Waitlist Control
Started | 15 | 15
Completed | 10 | 11
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Waitlist Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (7.8) | 37.9 (9.6) | 37.3 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 13 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Positive Psychology (PP) Intervention
Description: Percentage of subjects who completed at least four of the five PP exercises.
Time Frame: Five weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 15 | 15
Participants | 10 | 11

2. Secondary Outcome: Subject Ratings of Ease of Completion of PP Exercises
Description: Measured by averaging the weekly 0-10 post-exercise Likert scale ratings of ease of completion of PP exercises provided by subjects with 0 being very difficult to complete and 10 being very easy to complete.
Time Frame: Five weeks
Population: Data were included from all participants who completed each exercise, even if the participant did not complete at least four of the five PP exercises required to demonstrate feasibility.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 12 | 11
score on a scale | 7.2 [6.2 to 8.0] | 7.5 [6.6 to 8.4]

3. Secondary Outcome: Subject Ratings of Utility of PP Exercises
Description: Measured by averaging the weekly 0-10 post-exercise Likert scale ratings of utility of PP exercises provided by subjects, with 0 being not helpful and 10 being very helpful.
Time Frame: Five weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 12 | 11
score on a scale | 7.1 [6.2 to 7.9] | 7.9 [7.3 to 8.6]

4. Secondary Outcome: Changes in Affect From Baseline to Five Weeks
Description: Measured by the Positive and Negative Affect Schedule (PANAS). PANAS is comprised of two 10-item mood scales, one measuring positive affect and the other measuring negative affect. Scores on the positive affect scale range form 10-50. Higher scores are associated with greater positive affect. Scores on the negative affect scale range from 10-50, with lower scores representing lower levels of negative affect.
Time Frame: Five weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 10 | 11
score on a scale
  Changes in PANAS Positive Affect | 4.75 [1.77 to 7.72] | -1.93 [-4.75 to 0.89]
  Changes in PANAS Negative Affect | -2.47 [-5.34 to 0.4] | 0.74 [-1.74 to 3.23]

5. Secondary Outcome: Changes in Trait Optimism From Baseline to Five Weeks
Description: Measured by the Life Orientation Test - Revised (LOT-R). Lot-R is a 6-item measure of trait optimism and pessimism. Scores range from 0-24. Higher scores are associated with greater optimism.
Time Frame: Five weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 10 | 11
score on a scale | 1.77 [0.06 to 3.48] | -1.26 [-2.76 to 0.24]

6. Secondary Outcome: Changes in Physical, Mental and Social Health From Baseline to Five Weeks
Description: Measured by Neuro-QoL. Neuro-QoL uses computer adaptive testing to assess 11 domains of physical, mental and social health including Ability to participate in Social Roles and Activities, Anxiety, Cognitive Function, Depression, Emotional and Behavioral Dyscontrol, Fatigue, Lower Extremity Function, Positive Affect and Well-being, Satisfaction with Social Roles and Activities, Stigma and Upper Extremity Function. Neuro-QoL generates T scores with a mean of 50 and standard deviation (SD) of 10, based on the norming sample used, for each domain. All Neuro-QoL domains are scored such that a high score reflects more of what is being measured.
Time Frame: Five weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 10 | 11
score on a scale
  Changes in Neuro-QoL Ability to Participate in Social Roles | 2.41 [-0.9 to 5.71] | 0.62 [-2.39 to 3.63]
  Changes in Neuro-QoL Cognitive Function | 0.82 [-2.05 to 3.7] | 4.45 [1.93 to 6.97]
  Changes in Neuro-QoL Lower Extremity Function | 1.3 [-0.72 to 3.31] | -1.4 [-3.25 to 0.44]
  Changes in Neuro-QoL Positive Affect | 1.01 [-1.16 to 3.18] | -0.85 [-2.77 to 1.07]
  Changes in Neuro-QoL Satisfaction with Social Roles | 3.42 [0.37 to 6.47] | 0.52 [-2.24 to 3.27]
  Changes in Neur-QoL Upper Extremity Function | 1.71 [-0.72 to 4.13] | -1.28 [-3.42 to 0.86]
  Changes in Neuro-QoL Anxiety | -1.62 [-4.95 to 1.71] | -0.66 [-3.58 to 2.27]
  Changes in Neuro-QoL Depression | -1.46 [-3.97 to 1.04] | 0.02 [-2.19 to 2.22]
  Changes in Neuro-QoL Emotional and Behavioral Dyscontrol | -3.27 [-7.89 to 1.35] | -0.96 [-5.17 to 3.25]
  Changes in Neuro-QoL Fatigue | -2.22 [-5.13 to 0.69] | 0.4 [-2.29 to 3.09]
  Changes in Neuro-QoL Stigma | -1.48 [-3.8 to 0.83] | -1.47 [-3.5 to 0.57]

7. Secondary Outcome: Changes in Resilience From Baseline to Five Weeks
Description: Measured by the Brief Resilience Scale (BRS). BRS is a 6-item measure of resilience with scores ranging from 1-5. Higher scores are associated with greater resilience.
Time Frame: Five weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 10 | 11
score on a scale | 0.2 [-0.1 to 0.49] | 0.21 [-0.06 to 0.48]

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: It does not differ from the clinicaltrials.gov definition.
Groups:
- Waitlist Control - No Intervention; Waitlist Control - Intervention: Subjects randomized to the waitlist control group will complete study questionnaires at enrollment, Week 5 and Week 10. They will also complete 5 weeks of PP exercises, one exercise per week, during the extension phase (weeks 6-10) of the study.
  Positive psychology: 5-week positive psychology intervention
Arm/Group | Intervention | Waitlist Control - No Intervention | Waitlist Control - Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
This study had a small sample size and numerous outcome measures. This may have limited our ability to see statistically significant changes across broader health-related quality of life outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT06891937/Prot_SAP_000.pdf